CLINICAL TRIAL: NCT03516188
Title: Open-label Antacid-controlled Randomized Study on Effectiveness of Alginate-antacid Preparation (Gaviscon-Advance®) in Suppression of Post-supper Acid-pocket, Night-time Acid-reflux and Symptoms in Obese Participants
Brief Title: Efficacy of Gaviscon-Advance® in Suppressing Post-supper Acid-pocket and Night-time Acid-reflux in Obese Participants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Yeong Yeh Lee, Professor Dr, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15020071
Record Dates: First submitted 2017-10-18; First posted 2018-05-04 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Gastroesophageal Reflux Disease; Acid Reflux; Obesity
Keywords: Gastroesophageal Reflux Disease; Acid pocket; Acid Reflux; Alginate antacid; Obesity
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity

STUDY DESIGN:
Intervention Model Description: Asymptomatic obese patients will be randomised into either groups according to alginate antacid group [Gaviscon Advance (GA), Reckitt Benckiser, UK] and non antacid alginate group [simple antacid]. Both groups will be studied for 48 hours using the ambulatory wireless capsule and pH impedance. Participants according to their group will take either alginate antcid [Gaviscon Advance (GA), Reckitt Benckiser, UK] or non alginate antacid [simple antacid] which has equivalent strength of antacid after taking late night standardised meals.
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alginate-antacid group (Experimental): Participants will take normal meals with late night supper (i.e.two chicken burgers and one cup or 250 ml of teh-tarik) plus alginate-antacid.
  Interventions: Drug: Alginate-antacid group
- Non antacid alginate group (Experimental): Participants will take normal meals with late night supper (i.e.two chicken burgers and one cup or 250 ml of teh-tarik) plus antacid alone.
  Interventions: Drug: Non antacid alginate group

INTERVENTIONS:
Drug: Alginate-antacid group — Participants will be given 10 mL of alginate-antacid preparation (Gaviscon-Advance®, Reckitt-Benckiser, United Kingdom)
  Other Names: Gaviscon-Advance®
  Arms: Alginate-antacid group
Drug: Non antacid alginate group — Participants will be given 4 mL of magnesium tri-silicate which has equivalent strength and component with Gaviscon-Advance® except it is alginate-free.
  Other Names: Magnesium tri-silicate
  Arms: Non antacid alginate group

SUMMARY:
A randomized, open-label study with antacid-control will be performed over 48 hours period by continuous pH impedance and bravo capsule monitoring. Asymptomatic obese patients will be separated into either groups according to alginate antacid group [Gaviscon Advance (GA)®, Reckitt Benckiser, UK] and non antacid alginate group [simple antacid]. Both groups will be studied for 48 hours using the ambulatory wireless capsule and pH impedance. Participants according to their group will take either alginate antcid [Gaviscon Advance (GA)®, Reckitt Benckiser, UK] or non alginate antacid [simple antacid] which has equivalent strength of antacid after taking late night standardised meals.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) with symptoms of heartburn and acid regurgitation is a common disorder especially in overweight and obese persons who are at increased risk for GERD. Late night supper, an usual eating habit in many parts of the world, may worsen GERD and especially so among the obese, and this may be due to increased reflux from acid pocket.

Acid pocket in the proximal part of stomach after meals has been shown to be an important mechanism of GERD. The acid pocket is increasingly recognized as a source from which acid reflux events originate. To what extent changes in acidity of the acid pocket contribute to the therapeutic effect of alginate antacid formulation is inconsistent. The other findings suggested that the main mechanism of action for the alginate-antacid combination is to displace the post-prandial acid pocket rather than mechanically containing it.

Therefore, the outcomes of the study will allow us to determine whether late night supper worsen acid pocket, night time reflux and symptoms and whether an alginate antacid preparation (Gaviscon Advance®) is useful in suppression of acid pocket, night time refluxes and symptom (s). A benefit is that this study may inform doctors and advise participants of GERD side-effects of late night supper and how Gaviscon Advance may help.

ELIGIBILITY:
Inclusion Criteria:

1. Aged greater than or equal to 18 years and less than or equal to 70 years.
2. BMI >27.5 (based on kg/m2)

4. Not taking acid suppressant PPI and H2 receptor blockers 5. Not taking antacids or alginate preparations, except those administered as part of study procedure.

Exclusion Criteria:

1. Those with gastrointestinal symptoms indicative of GERD, gastric carcinoma, previous or current peptic ulcer disease.
2. Those with a history of upper GI surgery prior to this.
3. Those with haematological disorders, bleeding tendency, recurrent nose bleeds or treatment with anti-coagulants).
4. Those who had any previous history of allergy or known intolerance to any of the study drugs or the following formulation constituents: Gaviscon® liquid: sodium alginate, sodium bicarbonate and calcium carbonate
5. Those with physical, neurological or psychiatric conditions preventing repeated visits to hospital or compliance with study procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Duration of acid-pocket | 48 hours
  Duration of acid-pocket will be assessed using Bravo capsules. The unit of measure is in minutes.

SECONDARY OUTCOMES:
Symptom response | 48 hours
  Symptom response will be assessed using visual analogue scale (0 - 10).
Acidity of acid-pocket | 48 hours
  Acidity of acid-pocket will be assessed using Bravo capsules. The unit of measure is in pH.
Frequency of night-time reflux | 48 hours
  Frequency of night-time reflux will be assessed using pH-impedance studies.

CONTACTS AND LOCATIONS:
Overall Officials: Yeong Yeh Lee, MD, PhD, Principal Investigator — Universiti Sains Malaysia
Locations (1):
- Hospitial Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

REFERENCES:
- [Derived] Deraman MA, Abdul Hafidz MI, Lawenko RM, Ma ZF, Wong MS, Coyle C, Lee YY. Randomised clinical trial: the effectiveness of Gaviscon Advance vs non-alginate antacid in suppression of acid pocket and post-prandial reflux in obese individuals after late-night supper. Aliment Pharmacol Ther. 2020 Jun;51(11):1014-1021. doi: 10.1111/apt.15746. Epub 2020 Apr 28. PMID 32343001